CLINICAL TRIAL: NCT00934856
Title: An Open-Label, Multi-Center Phase I/II Study of the Safety and Tolerability of the Combination of Trastuzumab-MCC-DM1 (T-DM1) With Docetaxel, and Potentially Pertuzumab, for Treatment for Patients With Advanced Breast Cancer
Brief Title: A Study of Trastuzumab Emtansine (T-DM1) in Combination With Docetaxel, and Potentially Pertuzumab, in Participants With Advanced Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BP22572; 2009-010000-28 (EudraCT Number)
Record Dates: First submitted 2009-07-06; First posted 2009-07-08 (Estimated); Results first posted 2017-04-06 (Actual); Last update posted 2017-04-06 (Actual); Status verified 2017-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; pertuzumab; Ado-Trastuzumab Emtansine

ARMS (6):
- MBC: T-DM1 2.4 mg/kg + Doc 75 mg/m^2 (over 2 days) (Experimental): Participants with human epidermal growth factor receptor 2 (HER2)-positive MBC will receive docetaxel (Doc) 75 milligrams per square meter (mg/m^2) intravenous (IV) infusion on Day 1 and T-DM1 2.4 milligrams per kilogram (mg/kg) IV infusion on Day 2 of Cycle 1 followed by T-DM1 75 mg/m^2 and docetaxel 2.4 mg/kg IV infusion on Day 1 of each 3-week cycle for a minimum of 6 cycles. After 6 cycles, docetaxel 75 mg/m^2 will be stopped and T-DM1 2.4 mg/kg will be continued until confirmed evidence of disease progression, unacceptable toxicity, or withdrawal of participant consent.
  Interventions: Drug: Docetaxel; Drug: Trastuzumab emtansine
- MBC: T-DM1 2.4 mg/kg + Doc 60 mg/m^2 (over 2 days) (Experimental): Participants with HER2-positive MBC will receive docetaxel 60 mg/m^2 IV infusion on Day 1 and T-DM1 2.4 mg/kg IV infusion on Day 2 of Cycle 1 followed by T-DM1 60 mg/m^2 and docetaxel 2.4 mg/kg IV infusion on Day 1 of each 3-week cycle for a minimum of 6 cycles. After 6 cycles, docetaxel 60 mg/m^2 will be stopped and T-DM1 2.4 mg/kg will be continued until confirmed evidence of disease progression, unacceptable toxicity, or withdrawal of participant consent.
  Interventions: Drug: Docetaxel; Drug: Trastuzumab emtansine
- MBC: T-DM1 2.4 mg/kg + Doc 60 mg/m^2 (same day) (Experimental): Participants with HER2-positive MBC will receive docetaxel 60 mg/m^2 IV infusion and T-DM1 2.4 mg/kg IV infusion on Day 1 of each 3-week cycle for a minimum of 6 cycles. After 6 cycles, docetaxel 60 mg/m^2 will be stopped and T-DM1 2.4 mg/kg will be continued until confirmed evidence of disease progression, unacceptable toxicity, or withdrawal of participant consent.
  Interventions: Drug: Docetaxel; Drug: Trastuzumab emtansine
- MBC: T-DM1 3.6 mg/kg + Doc 60 mg/m^2 (same day) (Experimental): Participants with HER2-positive MBC will receive docetaxel 60 mg/m^2 IV infusion and T-DM1 3.6 mg/kg IV infusion on Day 1 of each 3-week cycle for a minimum of 6 cycles. After 6 cycles, docetaxel 60 mg/m^2 will be stopped and T-DM1 3.6 mg/kg will be continued until confirmed evidence of disease progression, unacceptable toxicity, or withdrawal of participant consent.
  Interventions: Drug: Docetaxel; Drug: Trastuzumab emtansine
- LABC: T-DM1 + Doc (Doublet Regimen) (Experimental): Participants with HER2-positive LABC will receive T-DM1 3.6 mg/kg IV infusion and docetaxel 60/75/100 mg/m^2 IV infusion on Day 1 of each 3-week cycle, for 6 cycles. Study treatment will be administered for up to 6 cycles or until unacceptable toxicity, and prior to surgery.
  Interventions: Drug: Docetaxel; Drug: Trastuzumab emtansine
- LABC: T-DM1 + Doc + Pertuzumab (Triplet Regimen) (Experimental): Participants with HER2-positive LABC will receive T-DM1 3.6 mg/kg Iv infusion, docetaxel 60/75 mg/m^2 IV infusion, and pertuzumab 840 mg (for Cycle 1) or 420 mg (for remaining cycles) IV infusion on Day 1 of each 3-week cycle, for 6 cycles. Study treatment will be administered for up to 6 cycles or until unacceptable toxicity, and prior to surgery.
  Interventions: Drug: Docetaxel; Drug: Pertuzumab; Drug: Trastuzumab emtansine

INTERVENTIONS:
Drug: Docetaxel — Docetaxel will be administered on Day 1 of each 3-week cycle at a dose specified in the respective arms (as per summary of product characteristics [SmPC]).
Drug: Pertuzumab — Pertuzumab at a loading dose of 840 mg IV infusion on Day 1 of Cycle 1 followed by maintenance dose of 420 mg IV infusion on Day 1 of each 3-week cycle.
  Arms: LABC: T-DM1 + Doc + Pertuzumab (Triplet Regimen)
Drug: Trastuzumab emtansine — T-DM1 will be administered on Day 1 or Day 2 of each 3-week cycle at a dose specified in the respective arms.
  Other Names: T-DM1

SUMMARY:
This is an open-label, multi-center, non-randomized study of the safety and tolerability of the combination of T-DM1 plus docetaxel for the treatment of participants with metastatic breast cancer (MBC) and of T-DM1 plus docetaxel with or without pertuzumab, for the treatment of participants with locally advanced breast cancer (LABC). The study comprises an initial dose finding (feasibility) part to determine the maximum tolerated dose (MTD) of T-DM1 and docetaxel, followed by an extension part aiming to consolidate the safety and efficacy of the recommended docetaxel/T-DM1 combination regimen.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status 0-1 (ECOG performance status of 2 will be allowed if only due to debilitating bone disease)
* HER2-positive metastatic or locally advanced breast cancer

For MBC participants:

* Documented metastatic or inoperable locally advanced (without meeting LABC criteria) disease, amenable for treatment with docetaxel
* History of disease progression within 3 months prior to study entry

For LABC participants:

* Newly diagnosed locally advanced breast cancer, Stage IIA-IIIC (American Joint Committee on Cancer [AJCC] staging system)

Exclusion Criteria:

* Significant cardiac disease
* Inadequate bone marrow, liver or renal function

For MBC participants:

* Participants must not have received radiotherapy for the treatment of metastatic or locally recurrent/advanced disease other than for the relief of pain in progressing metastatic bone lesions and/or brain metastases
* Brain metastases that are untreated, symptomatic or require therapy to control symptoms; or any radiation, surgery, or other therapy to control symptoms from brain metastasis within 2 months of the first study treatment.

For LABC participants:

* Clinically or radiologically detectable metastasis (M1 disease)
* Participants for whom surgery as primary intent procedure is the best option to treat their disease
* Participants must not have received any systemic or loco-regional anti-cancer therapy for the treatment of locally advanced disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2009-07 (Actual); Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (7):
- United States (2):
  - Charlotte, North Carolina
  - Houston, Texas
- France (2):
  - Dijon
  - Saint-Herblain
- Spain (2):
  - Barcelona, Barcelona
  - Madrid, Madrid
- Dundee, United Kingdom

REFERENCES:
- [Derived] Martin M, Fumoleau P, Dewar JA, Albanell J, Limentani SA, Campone M, Chang JC, Patre M, Strasak A, de Haas SL, Xu J, Garcia-Saenz JA. Trastuzumab emtansine (T-DM1) plus docetaxel with or without pertuzumab in patients with HER2-positive locally advanced or metastatic breast cancer: results from a phase Ib/IIa study. Ann Oncol. 2016 Jul;27(7):1249-56. doi: 10.1093/annonc/mdw157. Epub 2016 Apr 6. PMID 27052654

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Overall 152 participants were screened, of which 98 participants were enrolled (25 participants with metastatic breast cancer [MBC] and 73 participants with locally advanced breast cancer [LABC]) and included in the study.
Groups:
- MBC: T-DM1 2.4 mg/kg + Doc 75 mg/m^2 (Over 2 Days): Feasibility part: Participants with human epidermal growth factor receptor 2 (HER2)-positive MBC received docetaxel (Doc) 75 milligrams per square meter (mg/m^2) intravenous (IV) infusion on Day 1 and trastuzumab emtansine (T-DM1) 2.4 milligrams per kilogram (mg/kg) IV infusion on Day 2 of Cycle 1 followed by T-DM1 75 mg/m^2 and docetaxel 2.4 mg/kg IV infusion on Day 1 of each 3-week cycle for a minimum of 6 cycles. After 6 cycles, docetaxel 75 mg/m^2 was stopped and T-DM1 2.4 mg/kg was continued until confirmed evidence of disease progression, unacceptable toxicity, or withdrawal of participant consent.
- MBC: T-DM1 2.4 mg/kg + Doc 60 mg/m^2 (Over 2 Days): Feasibility part: Participants with HER2-positive MBC received docetaxel 60 mg/m^2 IV infusion on Day 1 and T-DM1 2.4 mg/kg IV infusion on Day 2 of Cycle 1 followed by T-DM1 60 mg/m^2 and docetaxel 2.4 mg/kg IV infusion on Day 1 of each 3-week cycle for a minimum of 6 cycles. After 6 cycles, docetaxel 60 mg/m^2 was stopped and T-DM1 2.4 mg/kg was continued until confirmed evidence of disease progression, unacceptable toxicity, or withdrawal of participant consent.
- MBC: T-DM1 2.4 mg/kg + Doc 60 mg/m^2 (Same Day): Feasibility part: Participants with HER2-positive MBC received docetaxel 60 mg/m^2 IV infusion and T-DM1 2.4 mg/kg IV infusion on Day 1 of each 3-week cycle for a minimum of 6 cycles. After 6 cycles, docetaxel 60 mg/m^2 was stopped and T-DM1 2.4 mg/kg was continued until confirmed evidence of disease progression, unacceptable toxicity, or withdrawal of participant consent.
- MBC: T-DM1 3.6 mg/kg + Doc 60 mg/m^2 (Same Day): Feasibility and extension part: Participants with HER2-positive MBC received docetaxel 60 mg/m^2 IV infusion and T-DM1 3.6 mg/kg IV infusion on Day 1 of each 3-week cycle for a minimum of 6 cycles. After 6 cycles, docetaxel 60 mg/m^2 was stopped and T-DM1 3.6 mg/kg was continued until confirmed evidence of disease progression, unacceptable toxicity, or withdrawal of participant consent.
- LABC: T-DM1 + Doc (Doublet Regimen): Feasibility and extension part: Participants with HER2-positive LABC received T-DM1 3.6 mg/kg IV infusion and docetaxel 60/75/100 mg/m^2 IV infusion on Day 1 of each 3-week cycle, for 6 cycles. Study treatment was administered for up to 6 cycles or until unacceptable toxicity, and prior to surgery.
- LABC: T-DM1 + Doc + Pertuzumab (Triplet Regimen): Feasibility and extension part: Participants with HER2-positive LABC received T-DM1 3.6 mg/kg Iv infusion, docetaxel 60/75 mg/m^2 IV infusion, and pertuzumab 840 mg (for Cycle 1) or 420 mg (for remaining cycles) IV infusion on Day 1 of each 3-week cycle, for 6 cycles. Study treatment was administered for up to 6 cycles or until unacceptable toxicity, and prior to surgery.
Period: Feasibility Part
Arm/Group | MBC: T-DM1 2.4 mg/kg + Doc 75 mg/m^2 (Over 2 Days) | MBC: T-DM1 2.4 mg/kg + Doc 60 mg/m^2 (Over 2 Days) | MBC: T-DM1 2.4 mg/kg + Doc 60 mg/m^2 (Same Day) | MBC: T-DM1 3.6 mg/kg + Doc 60 mg/m^2 (Same Day) | LABC: T-DM1 + Doc (Doublet Regimen) | LABC: T-DM1 + Doc + Pertuzumab (Triplet Regimen)
Started | 6 | 6 | 3 | 6 | 12 | 9
Completed | 1 | 1 | 0 | 1 | 12 | 6
Not Completed | 5 | 5 | 3 | 5 | 0 | 3
Not completed — Progressive disease | 4 | 4 | 2 | 3 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 0 | 1 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 1
Period: Extension Part
Arm/Group | MBC: T-DM1 2.4 mg/kg + Doc 75 mg/m^2 (Over 2 Days) | MBC: T-DM1 2.4 mg/kg + Doc 60 mg/m^2 (Over 2 Days) | MBC: T-DM1 2.4 mg/kg + Doc 60 mg/m^2 (Same Day) | MBC: T-DM1 3.6 mg/kg + Doc 60 mg/m^2 (Same Day) | LABC: T-DM1 + Doc (Doublet Regimen) | LABC: T-DM1 + Doc + Pertuzumab (Triplet Regimen)
Started | 0 | 0 | 0 | 4 (New participants were enrolled in the extension part.) | 28 (New participants were enrolled in the extension part.) | 24 (New participants were enrolled in the extension part.)
Completed | 0 | 0 | 0 | 2 | 24 | 19
Not Completed | 0 | 0 | 0 | 2 | 4 | 5
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 4 | 4
Not completed — Progressive disease | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Non-compliance with drug | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study medication were included.
Groups:
- MBC: T-DM1 2.4 mg/kg + Doc 75 mg/m^2 (Over 2 Days): Feasibility part: Participants with HER2-positive MBC received docetaxel 75 mg/m^2 IV infusion on Day 1 and T-DM1 2.4 mg/kg IV infusion on Day 2 of Cycle 1 followed by T-DM1 75 mg/m^2 and docetaxel 2.4 mg/kg IV infusion on Day 1 of each 3-week cycle for a minimum of 6 cycles. After 6 cycles, docetaxel 75 mg/m^2 was stopped and T-DM1 2.4 mg/kg was continued until confirmed evidence of disease progression, unacceptable toxicity, or withdrawal of participant consent.
- Total: Total of all reporting groups
Arm/Group | MBC: T-DM1 2.4 mg/kg + Doc 75 mg/m^2 (Over 2 Days) | MBC: T-DM1 2.4 mg/kg + Doc 60 mg/m^2 (Over 2 Days) | MBC: T-DM1 2.4 mg/kg + Doc 60 mg/m^2 (Same Day) | MBC: T-DM1 3.6 mg/kg + Doc 60 mg/m^2 (Same Day) | LABC: T-DM1 + Doc (Doublet Regimen) | LABC: T-DM1 + Doc + Pertuzumab (Triplet Regimen) | Total
Number analyzed (Participants) | 6 | 6 | 3 | 10 | 40 | 33 | 98
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (7.16) | 50.7 (4.84) | 57 (12.12) | 48 (9.39) | 48.6 (9.73) | 54.2 (11.43) | 50.4 (10.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 3 | 10 | 40 | 33 | 98
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicity (DLT) - MBC and LABC Feasibility Population
Description: DLTs included (as per National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] grading): Grade 4 thrombocytopenia, thrombocytopenia of any grade with concurrent hemorrhage or requiring blood platelet transfusion, or thrombocytopenia not recovered by Day 21 to at least 100,000/microliter (mcL); Grade 4 neutropenia lasting for more than 7 days; Febrile neutropenia; Grade greater than or equal to (>/=) 3 neurotoxicity in the form of peripheral neuropathy or peripheral neurotoxicity not improving to baseline or Grade less than or equal to (</=) 1 by Day 21; Any non-hematological toxicity of Grade >/= 3 except for alopecia, fever, and chills, not improving to baseline or Grade </=1 by Day 21, despite adequate toxicity management; Any subjective intolerable toxicity felt by the investigator to be related to either study treatment; Any other treatment-related toxicity prohibiting the start of the Cycle 2 on Day 22; Fulminant skin rash.
Time Frame: Cycle 1 (up to 21 days)
Population: MBC and LABC feasibility population: All participants who received at least one dose of study medication and included in the feasibility part of the study.
Measure: Number; unit: participants
Groups:
- MBC: T-DM1 2.4 mg/kg + Doc 75 mg/m^2 (Over 2 Days): Participants with HER2-positive MBC received docetaxel 75 mg/m^2 IV infusion on Day 1 and T-DM1 2.4 mg/kg IV infusion on Day 2 of Cycle 1 followed by T-DM1 75 mg/m^2 and docetaxel 2.4 mg/kg IV infusion on Day 1 of each 3-week cycle for a minimum of 6 cycles. After 6 cycles, docetaxel 75 mg/m^2 was stopped and T-DM1 2.4 mg/kg was continued until confirmed evidence of disease progression, unacceptable toxicity, or withdrawal of participant consent.
- MBC: T-DM1 2.4 mg/kg + Doc 60 mg/m^2 (Over 2 Days): Participants with HER2-positive MBC received docetaxel 60 mg/m^2 IV infusion on Day 1 and T-DM1 2.4 mg/kg IV infusion on Day 2 of Cycle 1 followed by T-DM1 60 mg/m^2 and docetaxel 2.4 mg/kg IV infusion on Day 1 of each 3-week cycle for a minimum of 6 cycles. After 6 cycles, docetaxel 60 mg/m^2 was stopped and T-DM1 2.4 mg/kg was continued until confirmed evidence of disease progression, unacceptable toxicity, or withdrawal of participant consent.
- MBC: T-DM1 2.4 mg/kg + Doc 60 mg/m^2 (Same Day): Participants with HER2-positive MBC received docetaxel 60 mg/m^2 IV infusion and T-DM1 2.4 mg/kg IV infusion on Day 1 of each 3-week cycle for a minimum of 6 cycles. After 6 cycles, docetaxel 60 mg/m^2 was stopped and T-DM1 2.4 mg/kg was continued until confirmed evidence of disease progression, unacceptable toxicity, or withdrawal of participant consent.
- MBC: T-DM1 3.6 mg/kg + Doc 60 mg/m^2 (Same Day): Participants with HER2-positive MBC received docetaxel 60 mg/m^2 IV infusion and T-DM1 3.6 mg/kg IV infusion on Day 1 of each 3-week cycle for a minimum of 6 cycles. After 6 cycles, docetaxel 60 mg/m^2 was stopped and T-DM1 3.6 mg/kg was continued until confirmed evidence of disease progression, unacceptable toxicity, or withdrawal of participant consent.
- LABC: T-DM1 + Doc (Doublet Regimen): Participants with HER2-positive LABC received T-DM1 3.6 mg/kg IV infusion and docetaxel 60/75/100 mg/m^2 IV infusion on Day 1 of each 3-week cycle, for 6 cycles. Study treatment was administered for up to 6 cycles or until unacceptable toxicity, and prior to surgery.
- LABC: T-DM1 + Doc + Pertuzumab (Triplet Regimen): Participants with HER2-positive LABC received T-DM1 3.6 mg/kg Iv infusion, docetaxel 60/75 mg/m^2 IV infusion, and pertuzumab 840 mg (for Cycle 1) or 420 mg (for remaining cycles) IV infusion on Day 1 of each 3-week cycle, for 6 cycles. Study treatment was administered for up to 6 cycles or until unacceptable toxicity, and prior to surgery.
Arm/Group | MBC: T-DM1 2.4 mg/kg + Doc 75 mg/m^2 (Over 2 Days) | MBC: T-DM1 2.4 mg/kg + Doc 60 mg/m^2 (Over 2 Days) | MBC: T-DM1 2.4 mg/kg + Doc 60 mg/m^2 (Same Day) | MBC: T-DM1 3.6 mg/kg + Doc 60 mg/m^2 (Same Day) | LABC: T-DM1 + Doc (Doublet Regimen) | LABC: T-DM1 + Doc + Pertuzumab (Triplet Regimen)
Number analyzed (Participants) | 6 | 6 | 3 | 6 | 12 | 9
participants | 2 | 1 | 0 | 1 | 2 | 2

2. Primary Outcome: Percentage of Participants With Adverse Events (AEs) or Serious AEs (SAEs) - MBC and LABC Population
Description: An AE is any new untoward medical occurrence or worsening of a pre-existing medical condition which does not necessarily have a causal relationship with this treatment. SAE is any untoward medical occurrence that at any dose results in death, is life-threatening, requires in-patient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, results in development of drug dependency or drug abuse, is an important medical event.
Time Frame: Baseline up to 28 days after last dose for MBC participants and for LABC participants who could not undergo surgery, and up to 6 weeks post-surgery for LABC participants who underwent surgery (maximum up to approximately 3 years)
Population: All participants who received at least one dose of study medication were included.
Measure: Number; unit: percentage of participants
Arm/Group | MBC: T-DM1 2.4 mg/kg + Doc 75 mg/m^2 (Over 2 Days) | MBC: T-DM1 2.4 mg/kg + Doc 60 mg/m^2 (Over 2 Days) | MBC: T-DM1 2.4 mg/kg + Doc 60 mg/m^2 (Same Day) | MBC: T-DM1 3.6 mg/kg + Doc 60 mg/m^2 (Same Day) | LABC: T-DM1 + Doc (Doublet Regimen) | LABC: T-DM1 + Doc + Pertuzumab (Triplet Regimen)
Number analyzed (Participants) | 6 | 6 | 3 | 10 | 40 | 33
percentage of participants
  AEs | 100 | 100 | 100 | 100 | 100 | 100
  SAEs | 33.3 | 33.3 | 66.7 | 40.0 | 22.5 | 27.3

3. Secondary Outcome: Percentage of Participants With Progression-Free Survival (PFS) Event - MBC Population
Description: PFS was defined as the time interval between the date of the start of treatment and the date of first documentation of progressive disease (PD) or death from any cause, whichever occurred first. Response was based on Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.0 (v1.0). For target lesions (TLs), PD was at least a 20 percent (%) increase in the sum of longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more lesions. For non-target lesions (NTLs), PD was the appearance of one or more new lesions and/or unequivocal progression of existing NTLs. Data for participants without PD or death was censored at the time of the last response assessment. Percentage of participants with PFS event was calculated as the (number of participants with PFS event [PD or death]) divided by (total number of participants), and then multiplied by 100.
Time Frame: Baseline until disease progression or death (up to approximately 3 years)
Population: MBC population: All participants with MBC who received at least one dose of study medication were included.
Measure: Number; unit: percentage of participants
Groups:
- Overall MBC Participants: Participants with MBC who were enrolled in the study and who received at least one dose of study medication
Arm/Group | Overall MBC Participants
Number analyzed (Participants) | 25
percentage of participants | 60.0

4. Secondary Outcome: PFS - MBC Population
Description: PFS was defined as the time interval between the date of the start of treatment and the date of first documentation of PD or death from any cause, whichever occurred first. Response was based on RECIST v1.0. For TLs, PD was at least a 20 % increase in the sum of LD of TLs, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more lesions. For NTLs, PD was the appearance of one or more new lesions and/or unequivocal progression of existing NTLs. Median PFS time was calculated using Kaplan-Meier estimates. Data for participants without PD or death was censored at the time of the last response assessment.
Time Frame: Baseline until disease progression or death (up to approximately 3 years)
Population: MBC population
Measure: Median (Full Range); unit: months
Arm/Group | Overall MBC Participants
Number analyzed (Participants) | 25
months | 13.8 [1.6 to 33.5]

5. Secondary Outcome: Percentage of Participants With a Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR) - MBC Population
Description: BOR was defined as CR or PR recorded from baseline until disease progression/recurrence according to RECIST v1.0 criteria. For TLs, CR was defined as the disappearance of all TLs, and PR was defined as at least a 30% decrease in the sum of LDs of the TLs, taking as a reference the baseline (BL) sum of LDs. For NTLs, CR was defined as the disappearance of all NTLs and normalization of tumor marker levels. Percentage of participants with BOR rate was calculated as the (number of participants with CR or PR) divided by (total number of participants), and then multiplied by 100. The 95% confidence interval (Cl) was determined using the Pearson-Clopper method.
Time Frame: Baseline until disease progression or recurrence (up to approximately 3 years)
Population: MBC population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Overall MBC Participants
Number analyzed (Participants) | 25
percentage of participants | 80.0 [59.3 to 93.2]

6. Secondary Outcome: Percentage of Participants With Treatment Failure - MBC Population
Description: Treatment failure was defined as the discontinuation of treatment for any reason, including the following qualifying events: PD, death from any cause, withdrawal from study treatment, or initiation of nonprotocol anti-cancer therapy. Percentage of participants with treatment failure was calculated as the (number of participants with treatment failure) divided by (total number of participants), and then multiplied by 100.
Time Frame: Baseline until end of treatment (up to 39.8 months)
Population: MBC population
Measure: Number; unit: percentage of participants
Arm/Group | Overall MBC Participants
Number analyzed (Participants) | 25
percentage of participants | 64.0

7. Secondary Outcome: Time to Treatment Failure (TTF) - MBC Population
Description: TTF was defined as the time interval between the date of start of treatment and the date of PD, death from any cause, withdrawal from study treatment, or initiation of non-protocol anti-cancer therapy, whichever occurred first. Participants without an event at the time of the analysis were censored at the date of the last follow-up assessment. Median TTF was estimated using the Kaplan-Meier method.
Time Frame: Baseline until end of treatment (up to 39.8 months)
Population: MBC population
Measure: Median (Full Range); unit: months
Arm/Group | Overall MBC Participants
Number analyzed (Participants) | 25
months | 13.8 [1.4 to 39.8]

8. Secondary Outcome: Percentage of Participants With CR or PR or Stable Disease (SD) for at Least 6 Months [Clinical Benefit Rate (CBR)] - MBC Population
Description: CBR was defined as percentage of participants experiencing SD of at least 6 months from the start of treatment plus CR or PR according to the RECIST v1.0 criteria. For TLs: CR- disappearance of all TLs. PR- at least 30% decrease in the sum of LDs of the TLs, taking as a reference the BL sum of LDs. PD- at least 20% increase in the sum of LD of TLs, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more lesions. SD- neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD. For NTLs: CR- disappearance of all NTLs and normalization of tumor marker levels. SD- persistence of one or more NTLs and/or maintenance of tumor marker level above the normal limits. Percentage of participants= number of participants with CR/PR/SD divided by total number of participants, and then multiplied by 100. 95% CI was determined using the Pearson-Clopper method.
Time Frame: Baseline until disease progression, recurrence or death (up to approximately 3 years)
Population: MBC population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Overall MBC Participants
Number analyzed (Participants) | 25
percentage of participants | 92.0 [74.0 to 99.0]

9. Secondary Outcome: Duration of Response - MBC Population
Description: Duration of response was calculated for participants with CR or PR based on the RECIST v1.0 criteria. Duration of response was defined as the time interval between the date the CR or PR was first recorded and the date on which PD was first noted or date of death, whichever occurred first. Participants with no documented PD after CR or PR were censored at the last date at which they were known to have had the CR or PR, respectively. Median duration of response was estimated using the Kaplan-Meier method.
Time Frame: Baseline until disease progression, recurrence or death (up to approximately 3 years)
Population: MBC population
Measure: Median (Full Range); unit: months
Arm/Group | Overall MBC Participants
Number analyzed (Participants) | 25
months | 12.4 [3.9 to 32.7]

10. Secondary Outcome: Percentage of Participants With Pathological CR (pCR) - LABC Population
Description: The pCR was defined as the absence of invasive neoplastic cells at microscopic examination of the tumor remnants and lymph nodes after surgery following primary systemic therapy.
Time Frame: Within 6 weeks of post-surgery (up to approximately 3 years)
Population: LABC population: All participants with LABC who received at least one dose of study medication.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LABC: T-DM1 + Doc (Doublet Regimen) | LABC: T-DM1 + Doc + Pertuzumab (Triplet Regimen)
Number analyzed (Participants) | 40 | 33
percentage of participants | 60.0 [43.3 to 75.1] | 60.6 [42.1 to 77.1]

11. Secondary Outcome: Percentage of Participants With a BOR of CR or PR - LABC Population
Description: BOR was defined as CR or PR recorded from baseline until disease progression/recurrence according to RECIST v1.0 criteria. For TLs, CR was defined as the disappearance of all TLs, and PR was defined as at least a 30% decrease in the sum of LDs of the TLs, taking as a reference the baseline (BL) sum of LDs. For NTLs, CR was defined as the disappearance of all NTLs and normalization of tumor marker levels. Percentage of participants with BOR rate was calculated as the (number of participants with CR or PR) divided by (total number of participants), and then multiplied by 100. The 95% Cl was determined using the Pearson-Clopper method.
Time Frame: Baseline until disease progression, recurrence or death (up to approximately 3 years)
Population: LABC population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LABC: T-DM1 + Doc (Doublet Regimen) | LABC: T-DM1 + Doc + Pertuzumab (Triplet Regimen)
Number analyzed (Participants) | 40 | 33
percentage of participants | 70.0 [53.5 to 83.4] | 51.5 [33.5 to 69.2]

12. Secondary Outcome: Number of Participants With Anti-Therapeutic Antibody (ATA) Response to Trastuzumab - MBC and LABC Population
Description: Number of participants with ATA response was reported. Data for this outcome measure was planned to be reported for overall MBC and LABC participants and not by individual treatment arms.
Time Frame: Baseline (Day 1 of Cycle 1), Post baseline (at first follow-up visit [28 days after last dose of study drug][up to approximately 145 weeks])
Population: All participants who received at least one dose of study medication were included. Here, number analyzed=participants evaluable for ATA at specified time-point.
Measure: Number; unit: participants
Groups:
- Overall MBC and LABC Participants: All enrolled participants who received at least one dose of study medication
Arm/Group | Overall MBC and LABC Participants
Number analyzed (Participants) | 98
participants
  Baseline: number analyzed (Participants) | 89
  Baseline | 3
  Post-baseline: number analyzed (Participants) | 79
  Post-baseline | 3

13. Secondary Outcome: Maximum Observed Concentration (Cmax) of Serum Trastuzumab Emtansine
Time Frame: Cycle 1: pre-dose (Hour [Hr] 0), 0.25, 4 hrs post end of infusion (EOI) of T-DM1 on Day 2; on Days 3 and 8. Cycle 2: pre-dose (Hr 0), 0.25, 4 hrs post EOI of T-DM1 on Day 1; on Day 8 (1 cycle = 21 days) (T-DM1 infusion duration = 1.5 hrs)
Population: Pharmacokinetic (PK) analysis population: PK-evaluable participants were defined as participants who received at least one dose of T-DM1 or docetaxel with at least one post-dose concentration data point. Number analyzed = participants evaluable for specified cycle for each arm.
Measure: Mean (Standard Deviation); unit: micrograms per milliliter (mcg/mL)
Groups:
- MBC: T-DM1 2.4 mg/kg: All MBC participants who received T-DM1 2.4 mg/kg IV infusion.
- MBC: T-DM1 3.6 mg/kg: All MBC participants who received T-DM1 3.6 mg/kg IV infusion.
- LABC: T-DM1 3.6 mg/kg: All LABC participants who received T-DM1 3.6 mg/kg IV infusion.
Arm/Group | MBC: T-DM1 2.4 mg/kg | MBC: T-DM1 3.6 mg/kg | LABC: T-DM1 3.6 mg/kg
Number analyzed (Participants) | 15 | 10 | 73
micrograms per milliliter (mcg/mL)
  Cycle 1 | 78.6 (16.6) | 76.2 (36.4) | 85.7 (15.3)
  Cycle 2: number analyzed (Participants) | 14 | 9 | 67
  Cycle 2 | 78.7 (16.7) | 93.7 (27.6) | 80.2 (18.4)

14. Secondary Outcome: Apparent Terminal Half-Life (t1/2) of Serum Trastuzumab Emtansine
Time Frame: Cycle 1: pre-dose (Hr 0), 0.25, 4 hrs post EOI of T-DM1 on Day 2; on Days 3 and 8. Cycle 2: pre-dose (Hr 0), 0.25, 4 hrs post EOI of T-DM1 on Day 1; on Day 8 (1 cycle = 21 days) (T-DM1 infusion duration = 1.5 hrs)
Population: PK analysis population. Overall number of participants analyzed = participants evaluable for this outcome measure. Number analyzed = participants evaluable for specified cycle for each arm.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | MBC: T-DM1 2.4 mg/kg | MBC: T-DM1 3.6 mg/kg | LABC: T-DM1 3.6 mg/kg
Number analyzed (Participants) | 15 | 8 | 72
days
  Cycle 1: number analyzed (Participants) | 15 | 7 | 72
  Cycle 1 | 2.79 (0.637) | 3.45 (0.779) | 3.46 (0.558)
  Cycle 2: number analyzed (Participants) | 14 | 8 | 63
  Cycle 2 | 3.14 (0.574) | 3.85 (0.568) | 3.62 (0.516)

15. Secondary Outcome: Area Under the Concentration-Time Curve From Time 0 to Infinity (AUCinf) of Serum Trastuzumab Emtansine
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: day*mcg/mL
Arm/Group | MBC: T-DM1 2.4 mg/kg | MBC: T-DM1 3.6 mg/kg | LABC: T-DM1 3.6 mg/kg
Number analyzed (Participants) | 15 | 8 | 72
day*mcg/mL
  Cycle 1: number analyzed (Participants) | 15 | 7 | 72
  Cycle 1 | 396 (124) | 447 (144) | 442 (90.7)
  Cycle 2: number analyzed (Participants) | 14 | 8 | 63
  Cycle 2 | 471 (94.5) | 556 (223) | 488 (123)

16. Secondary Outcome: Clearance (CL) of Serum Trastuzumab Emtansine
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: milliliters/day/kilogram (mL/day/kg)
Arm/Group | MBC: T-DM1 2.4 mg/kg | MBC: T-DM1 3.6 mg/kg | LABC: T-DM1 3.6 mg/kg
Number analyzed (Participants) | 15 | 8 | 72
milliliters/day/kilogram (mL/day/kg)
  Cycle 1: number analyzed (Participants) | 15 | 7 | 72
  Cycle 1 | 8.94 (12) | 8.87 (2.96) | 8.48 (1.86)
  Cycle 2: number analyzed (Participants) | 14 | 8 | 63
  Cycle 2 | 5.21 (1.27) | 7.16 (2.95) | 7.68 (2.73)

17. Secondary Outcome: Volume of Distribution at Steady State (Vss) of Serum Trastuzumab Emtansine
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | MBC: T-DM1 2.4 mg/kg | MBC: T-DM1 3.6 mg/kg | LABC: T-DM1 3.6 mg/kg
Number analyzed (Participants) | 15 | 8 | 72
mL/kg
  Cycle 1: number analyzed (Participants) | 15 | 7 | 72
  Cycle 1 | 22.1 (6.74) | 33.2 (9.13) | 33.2 (8.36)
  Cycle 2: number analyzed (Participants) | 14 | 8 | 63
  Cycle 2 | 17.7 (4.73) | 31.4 (16.9) | 28.8 (9.32)

18. Secondary Outcome: Cmax of Total Serum Trastuzumab
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | MBC: T-DM1 2.4 mg/kg | MBC: T-DM1 3.6 mg/kg | LABC: T-DM1 3.6 mg/kg
Number analyzed (Participants) | 15 | 10 | 73
mcg/mL
  Cycle 1 | 88.7 (22.6) | 89.2 (47.4) | 120 (46.6)
  Cycle 2: number analyzed (Participants) | 14 | 9 | 67
  Cycle 2 | 85.8 (17.5) | 97.7 (29.4) | 113 (43.8)

19. Secondary Outcome: t1/2 of Total Serum Trastuzumab
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: days
Arm/Group | MBC: T-DM1 2.4 mg/kg | MBC: T-DM1 3.6 mg/kg | LABC: T-DM1 3.6 mg/kg
Number analyzed (Participants) | 15 | 8 | 73
days
  Cycle 1: number analyzed (Participants) | 15 | 7 | 73
  Cycle 1 | 6.44 (2.6) | 6.38 (1.41) | 8.12 (4.2)
  Cycle 2: number analyzed (Participants) | 13 | 8 | 62
  Cycle 2 | 6.67 (1.92) | 7.83 (1.68) | 9.91 (5.01)

20. Secondary Outcome: AUCinf of Total Serum Trastuzumab
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: day*mcg/mL
Arm/Group | MBC: T-DM1 2.4 mg/kg | MBC: T-DM1 3.6 mg/kg | LABC: T-DM1 3.6 mg/kg
Number analyzed (Participants) | 15 | 8 | 73
day*mcg/mL
  Cycle 1: number analyzed (Participants) | 15 | 7 | 73
  Cycle 1 | 785 (429) | 707 (201) | 1210 (856)
  Cycle 2: number analyzed (Participants) | 13 | 8 | 62
  Cycle 2 | 809 (308) | 1040 (359) | 1570 (1180)

21. Secondary Outcome: CL of Total Serum Trastuzumab
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: mL/day/kg
Arm/Group | MBC: T-DM1 2.4 mg/kg | MBC: T-DM1 3.6 mg/kg | LABC: T-DM1 3.6 mg/kg
Number analyzed (Participants) | 15 | 8 | 73
mL/day/kg
  Cycle 1: number analyzed (Participants) | 15 | 7 | 73
  Cycle 1 | 6.78 (13.3) | 5.45 (1.46) | 4.22 (2.13)
  Cycle 2: number analyzed (Participants) | 13 | 8 | 62
  Cycle 2 | 3.32 (1.53) | 3.71 (1.23) | 3.38 (2.11)

22. Secondary Outcome: Vss of Total Serum Trastuzumab
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | MBC: T-DM1 2.4 mg/kg | MBC: T-DM1 3.6 mg/kg | LABC: T-DM1 3.6 mg/kg
Number analyzed (Participants) | 15 | 8 | 73
mL/kg
  Cycle 1: number analyzed (Participants) | 15 | 7 | 73
  Cycle 1 | 27 (7.16) | 41.3 (9.24) | 36.5 (12.7)
  Cycle 2: number analyzed (Participants) | 13 | 8 | 62
  Cycle 2 | 24.6 (5.05) | 36.4 (11.3) | 35.2 (12)

23. Secondary Outcome: Cmax of Plasma N2'-Deacetyl-N2'-(3-mercapto-1-oxopropyl)-Maytansine (DM1)
Description: DM1 is the metabolite of trastuzumab emtansine.
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | MBC: T-DM1 2.4 mg/kg | MBC: T-DM1 3.6 mg/kg | LABC: T-DM1 3.6 mg/kg
Number analyzed (Participants) | 13 | 9 | 73
nanograms per milliliter (ng/mL)
  Cycle 1 | 3.55 (1.6) | 3.42 (0.944) | 4.51 (1.38)
  Cycle 2: number analyzed (Participants) | 13 | 9 | 67
  Cycle 2 | 3.34 (0.815) | 3.9 (1.19) | 4.65 (1.57)

24. Secondary Outcome: t1/2 of Plasma DM1
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: days
Arm/Group | MBC: T-DM1 2.4 mg/kg | MBC: T-DM1 3.6 mg/kg | LABC: T-DM1 3.6 mg/kg
Number analyzed (Participants) | 12 | 7 | 68
days
  Cycle 1 | 1.12 (0.702) | 1.2 (0.985) | 1.87 (1.63)
  Cycle 2: number analyzed (Participants) | 2 | 1 | 31
  Cycle 2 | 3.75 (0.912) | 2.91 | 3.32 (0.7)

25. Secondary Outcome: AUCinf of Plasma DM1
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: day*ng/mL
Arm/Group | MBC: T-DM1 2.4 mg/kg | MBC: T-DM1 3.6 mg/kg | LABC: T-DM1 3.6 mg/kg
Number analyzed (Participants) | 12 | 7 | 68
day*ng/mL
  Cycle 1 | 5.72 (5.16) | 5.01 (2.54) | 9.38 (9.33)
  Cycle 2: number analyzed (Participants) | 2 | 1 | 31
  Cycle 2 | 17.8 (4.6) | 20 | 18.5 (4.28)

26. Secondary Outcome: Cmax of Plasma Docetaxel
Description: Docetaxel infusion duration = 1 hr (as per summary of product characteristics [SmPC])
Time Frame: Cycle 1: pre-dose (Hr 0), 0.25, 0.5, 1, 2, 4, 8, 23 hrs post EOI of docetaxel on Day 1. Cycle 2: pre-dose (Hr 0), 0.5 hr and 59 min after start of infusion, 0.25, 0.5, 1, 2, 4, 8, 23 hrs post EOI of docetaxel on Day 1 (1 cycle = 21 days)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- MBC: Docetaxel 75 mg/m^2: All MBC participants who received docetaxel 75 mg/m^2 IV infusion.
- MBC: Docetaxel 60 mg/m^2: All MBC participants who received docetaxel 60 mg/m^2 IV infusion.
- LABC: Docetaxel 60 mg/m^2: All LABC participants who received docetaxel 60 mg/m^2 IV infusion.
- LABC: Docetaxel 75 mg/m^2: All LABC participants who received docetaxel 75 mg/m^2 IV infusion.
- LABC: Docetaxel 100 mg/m^2: All LABC participants who received docetaxel 100 mg/m^2 IV infusion.
Arm/Group | MBC: Docetaxel 75 mg/m^2 | MBC: Docetaxel 60 mg/m^2 | LABC: Docetaxel 60 mg/m^2 | LABC: Docetaxel 75 mg/m^2 | LABC: Docetaxel 100 mg/m^2
Number analyzed (Participants) | 6 | 19 | 14 | 36 | 22
ng/mL
  Cycle 1 | 500 (216) | 1300 (829) | 1470 (551) | 1710 (426) | 2950 (1540)
  Cycle 2: number analyzed (Participants) | 6 | 17 | 12 | 35 | 19
  Cycle 2 | 791 (637) | 1320 (826) | 1590 (441) | 1960 (552) | 2790 (979)

27. Secondary Outcome: t1/2 of Plasma Docetaxel
Description: Docetaxel infusion duration = 1 hr (as per SmPC)
Time Frame: as for outcome 26
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: hours (hr)
Arm/Group | MBC: Docetaxel 75 mg/m^2 | MBC: Docetaxel 60 mg/m^2 | LABC: Docetaxel 60 mg/m^2 | LABC: Docetaxel 75 mg/m^2 | LABC: Docetaxel 100 mg/m^2
Number analyzed (Participants) | 6 | 19 | 14 | 36 | 22
hours (hr)
  Cycle 1 | 6.83 (4.22) | 5.17 (4.02) | 4.25 (5.61) | 8.29 (5.75) | 8.76 (3.82)
  Cycle 2: number analyzed (Participants) | 6 | 17 | 12 | 35 | 19
  Cycle 2 | 7.7 (4.15) | 7.88 (6.18) | 5.9 (3.83) | 6.69 (5.55) | 7.24 (3.58)

28. Secondary Outcome: AUCinf of Plasma Docetaxel
Description: Docetaxel infusion duration = 1 hr (as per SmPC)
Time Frame: as for outcome 26
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | MBC: Docetaxel 75 mg/m^2 | MBC: Docetaxel 60 mg/m^2 | LABC: Docetaxel 60 mg/m^2 | LABC: Docetaxel 75 mg/m^2 | LABC: Docetaxel 100 mg/m^2
Number analyzed (Participants) | 6 | 19 | 14 | 36 | 22
hr*ng/mL
  Cycle 1 | 1050 (475) | 1560 (874) | 1540 (421) | 2140 (669) | 4020 (2120)
  Cycle 2: number analyzed (Participants) | 6 | 17 | 12 | 35 | 19
  Cycle 2 | 1700 (1190) | 1710 (875) | 3260 (5100) | 2420 (887) | 3840 (1930)

29. Secondary Outcome: CL of Plasma Docetaxel
Description: Docetaxel infusion duration = 1 hr (as per SmPC)
Time Frame: as for outcome 26
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: liters/hour/square meter (L/hr/m^2)
Arm/Group | MBC: Docetaxel 75 mg/m^2 | MBC: Docetaxel 60 mg/m^2 | LABC: Docetaxel 60 mg/m^2 | LABC: Docetaxel 75 mg/m^2 | LABC: Docetaxel 100 mg/m^2
Number analyzed (Participants) | 6 | 19 | 14 | 36 | 22
liters/hour/square meter (L/hr/m^2)
  Cycle 1 | 82.2 (32.6) | 58.3 (40.9) | 42.8 (16.4) | 39.5 (16.8) | 30.5 (14.5)
  Cycle 2: number analyzed (Participants) | 6 | 17 | 12 | 35 | 19
  Cycle 2 | 59 (29.9) | 51.2 (38.5) | 32.6 (13.1) | 33.6 (11.9) | 27.9 (9.13)

30. Secondary Outcome: Vss of Plasma Docetaxel
Description: Docetaxel infusion duration = 1 hr (as per SmPC)
Time Frame: as for outcome 26
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: liters per square meter (L/m^2)
Arm/Group | MBC: Docetaxel 75 mg/m^2 | MBC: Docetaxel 60 mg/m^2 | LABC: Docetaxel 60 mg/m^2 | LABC: Docetaxel 75 mg/m^2 | LABC: Docetaxel 100 mg/m^2
Number analyzed (Participants) | 6 | 19 | 14 | 36 | 22
liters per square meter (L/m^2)
  Cycle 1 | 530 (398) | 203 (275) | 75 (113) | 126 (86.7) | 116 (73.3)
  Cycle 2: number analyzed (Participants) | 6 | 17 | 12 | 35 | 19
  Cycle 2 | 380 (257) | 253 (234) | 93.2 (64.7) | 79 (53.6) | 84.8 (39.1)

ADVERSE EVENTS:
Time Frame: Baseline up to 28 days after last dose for MBC participants and for LABC participants who could not undergo surgery, and up to 6 weeks post-surgery for LABC participants who underwent surgery (maximum up to approximately 3 years)
Description: All participants who received at least one dose of study medication were included.
Arm/Group | MBC: T-DM1 2.4 mg/kg + Doc 75 mg/m^2 (Over 2 Days) | MBC: T-DM1 2.4 mg/kg + Doc 60 mg/m^2 (Over 2 Days) | MBC: T-DM1 2.4 mg/kg + Doc 60 mg/m^2 (Same Day) | MBC: T-DM1 3.6 mg/kg + Doc 60 mg/m^2 (Same Day) | LABC: T-DM1 + Doc (Doublet Regimen) | LABC: T-DM1 + Doc + Pertuzumab (Triplet Regimen)
Serious Adverse Events (participants affected / at risk) | 2/6 | 2/6 | 2/3 | 4/10 | 9/40 | 9/33
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 3/3 | 10/10 | 40/40 | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MBC: T-DM1 2.4 mg/kg + Doc 75 mg/m^2 (Over 2 Days) (N=6) | MBC: T-DM1 2.4 mg/kg + Doc 60 mg/m^2 (Over 2 Days) (N=6) | MBC: T-DM1 2.4 mg/kg + Doc 60 mg/m^2 (Same Day) (N=3) | MBC: T-DM1 3.6 mg/kg + Doc 60 mg/m^2 (Same Day) (N=10) | LABC: T-DM1 + Doc (Doublet Regimen) (N=40) | LABC: T-DM1 + Doc + Pertuzumab (Triplet Regimen) (N=33)
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 2
Thrombosis in device (General disorders) | 1 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Uterine polyp (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 0 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hepatocellular injury (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0
Melanoderma (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dermatomyositis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 1
Anal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Device deployment issue (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MBC: T-DM1 2.4 mg/kg + Doc 75 mg/m^2 (Over 2 Days) (N=6) | MBC: T-DM1 2.4 mg/kg + Doc 60 mg/m^2 (Over 2 Days) (N=6) | MBC: T-DM1 2.4 mg/kg + Doc 60 mg/m^2 (Same Day) (N=3) | MBC: T-DM1 3.6 mg/kg + Doc 60 mg/m^2 (Same Day) (N=10) | LABC: T-DM1 + Doc (Doublet Regimen) (N=40) | LABC: T-DM1 + Doc + Pertuzumab (Triplet Regimen) (N=33)
Hot flush (Vascular disorders) | 0 | 1 | 0 | 0 | 5 | 0
Flushing (Vascular disorders) | 1 | 0 | 0 | 0 | 1 | 1
Haematoma (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pallor (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Varicose vein (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Tooth repair (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 6 | 5 | 1 | 6 | 25 | 20
Mucosal inflammation (General disorders) | 1 | 3 | 1 | 3 | 20 | 15
Pyrexia (General disorders) | 1 | 5 | 0 | 2 | 8 | 10
Fatigue (General disorders) | 0 | 1 | 1 | 1 | 10 | 9
Oedema peripheral (General disorders) | 0 | 1 | 0 | 2 | 3 | 1
Influenza like illness (General disorders) | 0 | 1 | 0 | 1 | 4 | 0
Chills (General disorders) | 0 | 2 | 1 | 0 | 1 | 1
Mucosal dryness (General disorders) | 0 | 0 | 0 | 0 | 1 | 3
Non-cardiac chest pain (General disorders) | 0 | 3 | 0 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 3 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 1
Feeling hot (General disorders) | 0 | 1 | 0 | 0 | 1 | 0
Axillary pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Local swelling (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Temperature intolerance (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Temperature regulation disorder (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Thrombosis in device (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vaccination site reaction (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 3 | 8 | 6
Anxiety (Psychiatric disorders) | 0 | 2 | 0 | 1 | 1 | 3
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 0
Metrorrhagia (Reproductive system and breast disorders) | 2 | 0 | 0 | 1 | 2 | 1
Menstruation irregular (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 4 | 1
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 1 | 1 | 1
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0 | 1 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 2 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Recall phenomenon (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Tooth avulsion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 0 | 1 | 11 | 7
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 0 | 1 | 8 | 4
Gamma-glutamyltransferase increased (Investigations) | 3 | 0 | 0 | 1 | 3 | 0
Blood lactate dehydrogenase increased (Investigations) | 2 | 0 | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 1 | 0 | 2 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Body temperature increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 1 | 0 | 0
Systolic dysfunction (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 1 | 6 | 21 | 19
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 0 | 4 | 4 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 2 | 4 | 4 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2 | 2 | 6
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 4 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 1 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 2 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 1
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Suffocation feeling (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 6 | 5 | 1 | 7 | 11 | 12
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 4 | 0 | 8 | 9 | 7
Leukopenia (Blood and lymphatic system disorders) | 5 | 3 | 1 | 4 | 3 | 3
Lymphopenia (Blood and lymphatic system disorders) | 5 | 1 | 0 | 3 | 3 | 4
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 3 | 4 | 4
Dysgeusia (Nervous system disorders) | 3 | 1 | 1 | 4 | 19 | 13
Headache (Nervous system disorders) | 2 | 1 | 1 | 4 | 12 | 11
Neuropathy peripheral (Nervous system disorders) | 2 | 3 | 1 | 2 | 8 | 5
Paraesthesia (Nervous system disorders) | 1 | 3 | 0 | 3 | 4 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 3 | 1
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 4 | 1
Dysaesthesia (Nervous system disorders) | 1 | 1 | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 1 | 0 | 1 | 0 | 0
Aphonia (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0
Burning sensation (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Sinus headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 1 | 2 | 1 | 4 | 15 | 16
Conjunctivitis (Eye disorders) | 0 | 2 | 1 | 1 | 6 | 2
Dry eye (Eye disorders) | 1 | 1 | 0 | 1 | 3 | 5
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0 | 6 | 2
Xerophthalmia (Eye disorders) | 0 | 0 | 0 | 0 | 2 | 2
Blepharospasm (Eye disorders) | 1 | 0 | 0 | 0 | 2 | 0
Conjunctival oedema (Eye disorders) | 0 | 0 | 0 | 0 | 2 | 1
Eye disorder (Eye disorders) | 0 | 0 | 0 | 0 | 3 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 1
Eye pain (Eye disorders) | 0 | 0 | 0 | 1 | 1 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 1 | 1 | 0
Visual acuity reduced (Eye disorders) | 1 | 0 | 0 | 0 | 1 | 0
Visual impairment (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 1
Dacryostenosis acquired (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0
Eyelids pruritus (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 2 | 1
Tinnitus (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 5 | 1 | 4 | 16 | 16
Diarrhoea (Gastrointestinal disorders) | 3 | 3 | 1 | 3 | 12 | 18
Constipation (Gastrointestinal disorders) | 1 | 1 | 3 | 3 | 19 | 11
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 2 | 3 | 14 | 10
Vomiting (Gastrointestinal disorders) | 1 | 2 | 1 | 5 | 11 | 11
Stomatitis (Gastrointestinal disorders) | 3 | 4 | 0 | 5 | 4 | 5
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 0 | 2 | 5 | 4
Abdominal pain upper (Gastrointestinal disorders) | 2 | 3 | 0 | 1 | 3 | 5
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 4 | 3
Odynophagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 5 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 3 | 3
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 4 | 3
Gingival bleeding (Gastrointestinal disorders) | 0 | 2 | 0 | 2 | 3 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 3 | 0 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 3 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 1
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 2
Aphthous Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Breath odour (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Epulis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Food poisoning (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Tooth loss (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hepatocellular injury (Hepatobiliary disorders) | 1 | 2 | 0 | 2 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1 | 5
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pyelocaliectasis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 4 | 0 | 4 | 20 | 12
Rash (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 8 | 11
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 8 | 4
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 9 | 3
Nail dystrophy (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 1 | 5 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 2 | 1 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 2 | 2
Eczema (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 1 | 1 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 3 | 1
Onychalgia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 1
Onycholysis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 2 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Madarosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 3 | 0 | 1 | 18 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 4 | 0 | 3 | 9 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 4 | 10 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 0 | 4 | 6 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0 | 0 | 6 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 3 | 4 | 3
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 1 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1 | 1 | 1
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 2 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2 | 1 | 2 | 9 | 9
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 2
Nasopharyngitis (Infections and infestations) | 3 | 0 | 1 | 5 | 7 | 1
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 3 | 4 | 3
Rhinitis (Infections and infestations) | 1 | 1 | 1 | 2 | 4 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 0 | 0 | 2 | 1
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 4 | 1
Influenza (Infections and infestations) | 1 | 1 | 0 | 0 | 3 | 0
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 0 | 2 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 2
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 1
Gingivitis (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 1
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 1
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 1
Cystitis (Infections and infestations) | 1 | 0 | 0 | 1 | 0 | 0
Eye infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2
Herpes zoster (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0
Hordeolum (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Device related infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Fungal skin infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Genital herpes (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Herpes virus infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Laryngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Mastitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Allodynia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.